CLINICAL TRIAL: NCT02324855
Title: Long Term Airway Clearance Therapy in Non Cystic Fibrosis Bronchiectasis: a Randomized Controlled Trial
Brief Title: Long-term Airway Clearance Therapy in Non-cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Exacerb_BQnoFQ
Record Dates: First submitted 2014-12-01; First posted 2014-12-24 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Bronchiectasis
Keywords: Autogenic drainage; Positive expiratory pressure; Airway clearance technique; Quality of life; Exacerbations; Chest physiotherapy
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): Subjects will receive the usual medical care in accordance with Spanish non cystic fibrosis bronchiectasis guidelines. In addition they will receive educational sessions about their disease and their pharmacology treatment.
- Chest physiotherapy plus usual care (Experimental): Subjects will introduce chest physiotherapy as part of their daily treatment
  Interventions: Other: Chest physiotherapy plus usual care

INTERVENTIONS:
Other: Chest physiotherapy plus usual care — Subjects will perform daily chest physiotherapy during at least 30 minutes. Patients will perform a slow expiratory airway clearance technique combined with positive expiratory pressure device (Acapella device, Murray et al.) Each patient will receive 12 supervised professional sessions (once a month).
  Arms: Chest physiotherapy plus usual care

SUMMARY:
The main aim is to analyze whether the routine use of chest physiotherapy in non cystic fibrosis bronchiectasis (NCFB) improves the cough severity and the quality of life in this population. In addition, the secondary end-points include incidences of exacerbations, changes in lung function, exercise capacity, airways inflammation, sputum analysis and eventual adverse events.

DETAILED DESCRIPTION:
The present project will be a single-blind , randomized, controlled trial of 12-month daily performing chest physiotherapy compared with usual care, followed by a 3-month intervention-free in non-cystic fibrosis bronchiectasis.

Intervention group will perform daily autonomous airway clearance techniques (positive expiratory pressure technique through Acapella device and autogenic drainage technique). Patients will receive professional sessions once a month.

Control group will receive their usual care and educational sessions about their disease. Physiotherapist will call them once a month.

During the study period the patients' pharmacological treatment remained unchanged

ELIGIBILITY:
Inclusion Criteria:

* Chronic sputum production during at least 3 months previous enrolment
* At least two confirmed exacerbations during the last year
* Patients able to understand how to perform the airway clearance techniques
* Clinically stable at time of study entry (defined as no requirement for antibiotics or change in respiratory medication in the preceding 4 wk)
* To be able to provide written, informed consent

Exclusion Criteria:

* Cystic Fibrosis
* Carry out regular chest physiotherapy.
* Active haemoptysis during the previous month or recurrent hemoptysis during the last year (more than 4 episodes)
* Waiting a pulmonary transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-10; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Cough severity (Auto-administered questionnaire: Leicester Cough Questionnaire) | 1 year
  Auto-administered questionnaire: Leicester Cough Questionnaire

SECONDARY OUTCOMES:
Quality of life (Quality of life-Bronchiectasis questionnaire) | 1 year
  Auto-administered questionaire: Quality of Life- Bronchiectasis
Exacerbation frequency | 1 year
  Number of exacerbation
Exercise capacity (Incremental field test: shuttle test) | 1 year
  Incremental field test: shuttle test
Lung function | 1 year
  Simple spirometry: Forced expiratory volume at 1 second, Forced vital capacity, Forced expiratory flow 25-75
Airway inflammation as assessed by spontaneous sputum analysis | 1 year
  Inflammatory sputum markers: Myeloperoxidase (MPO) and Cytokines (IL-8)

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Herrero, Msc, Principal Investigator — Universidad San Jorge
Locations (1):
- Universidad San Jorge, Zaragoza, Spain

REFERENCES:
- [Background] Murray MP, Pentland JL, Hill AT. A randomised crossover trial of chest physiotherapy in non-cystic fibrosis bronchiectasis. Eur Respir J. 2009 Nov;34(5):1086-92. doi: 10.1183/09031936.00055509. Epub 2009 Jun 18. PMID 19541717